CLINICAL TRIAL: NCT04419844
Title: Evaluation of TAR Technique in the Treatment of Huge Abdominal Wall Hernia and Large Abdominal Wall Defect With or Without Botox Injection .
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R.19.03.451 - 2019/03/11
Record Dates: First submitted 2020-06-03; First posted 2020-06-05 (Actual); Last update posted 2020-06-18 (Actual); Status verified 2020-05

CONDITIONS: TAR Technique
MeSH Terms: interventions — Tars; Botulinum Toxins, Type A

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TAR with Botox (Active Comparator): Evaluation of TAR technique in the treatment of huge abdominal wall hernia and large abdominal wall defect Botox injection .
  Interventions: Procedure: Tar with Botox
- TAR without Botox (Active Comparator): Evaluation of TAR technique in the treatment of huge abdominal wall hernia and large abdominal wall defect without Botox injection .
  Interventions: Procedure: Tar with Botox

INTERVENTIONS:
Procedure: Tar with Botox — Evaluation of TAR technique in the treatment of huge abdominal wall hernia and large abdominal wall defect with Botox injection .

SUMMARY:
Aim of the work In this study, we will evaluate posterior component separation (TAR) technique with or without Botox injection for open huge ventral hernia and large abdominal wall defect repair. The primary outcome will be recurrence while the secondary outcome will be infection, postoperative complications (bleeding and dehiscence), pain score, operative time, hospitalization, need for drain, time for drain removal and pulmonary function test before and after surgery.

This prospective clinical study will be performed on 40 eligible patients admitted to general surgery department at Mansoura University Hospi

ELIGIBILITY:
Inclusion Criteria:

* Adult patient fit for general anesthesia with huge ventral hernia (primary, incisional or recurrent).Any patient with large abdominal wall defect secondary to abdominal wall tumor excision or burst after surgery

Exclusion Criteria:

* Patients who are unfit for general anaesthesia. Poor pulmonary function tests. Pregnant females. Patient younger than 18 years. Immunodeficiency. Patient with psychiatric disease disabling surgical intervention. Patients who refuse to participate in our study.

Ages: 12 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-06-17 (Actual); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-06-02 (Estimated)

PRIMARY OUTCOMES:
Recurrence | one year
  Recurrence of the ventral hernia

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura University, Al Mansurah, Dakahlia Governorate, Egypt